CLINICAL TRIAL: NCT05863520
Title: A Comparison of Two School Based Interventions to Manage Anxiety in Autistic Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Emory University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-0521
Record Dates: First submitted 2023-03-14; First posted 2023-05-18 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder; Anxiety Disorders; Emotion Regulation
Keywords: intervention; schools; cognitive behavior therapy; group
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Up to 100 schools will be randomized to either Zones of Regulation or Facing Your Fears - School Based. Autistic students with anxiety within each school will be assigned to one of the programs.
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators will be masked to condition and collect post- intervention data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facing Your Fears - School Based (Active Comparator): Facing Your Fears-School Based (FYF-SB) is a 12 week school based group program comprised of psychoeducation (somatic management, development of positive self-statements and strategies for managing emotions), and graded exposure (facing fears a little at a time).
  Interventions: Behavioral: Facing Your Fears - School Based
- Zones of Regulation (Active Comparator): Zones of Regulation (ZOR) focuses on four different emotional states called "zones." Each zone is represented by different colors that represent different levels of emotions or arousal. ZOR includes psychoeducation about emotions and emotional states (e.g., reading facial expressions, identifying triggers for emotion dysregulations, using emotion regulation tools) and problem-solving strategies. In ZOR, students are also taught emotion regulation strategies (e.g., "calming", "cognitive" and "sensory" strategies) to stay in a specific zone and/or to move from one zone to another.
  Interventions: Behavioral: Zones of Regulation

INTERVENTIONS:
Behavioral: Zones of Regulation — ZOR is rooted in CBT principles and uses a metacognitive framework to increase awareness of feelings and to build regulation, prosocial skills, and overall wellness.
  Arms: Zones of Regulation
Behavioral: Facing Your Fears - School Based — FYF-SB is a CBT program for managing anxiety in autistic youth.
  Arms: Facing Your Fears - School Based

SUMMARY:
The goal of this clinical trial is to compare two school based interventions to manage anxiety in autistic students. The main question[s] it aims to answer are: 1) Compare the effectiveness of Facing Your Fears-School Based Program (FYF-SB) with Zones of Regulation (ZOR) on anxiety reduction and emotion regulation; and 2) examine the feasibility and satisfaction of FYF-SB and ZOR, according to students, caregivers and school providers. Autistic students with anxiety between 8-14 years will be randomized to either FYF-SB and ZOR. They will participate in one of the programs for 12 weeks and pre, post and follow-up measures will occur.

DETAILED DESCRIPTION:
Background and Significance: Anxiety is very common for autistic youth and can significantly limit functioning and full participation across settings. In school, anxiety may negatively impact students' attendance, school performance, peer relationships and extracurricular participation. Unfortunately, autistic youth have experienced long-standing difficulty accessing mental health care in community settings, and this difficulty is even more pronounced for youth from historically underserved racial and ethnic backgrounds. Cognitive-behavioral therapies (CBT) are evidence-based practices that are effective for anxious children with and without autism but have not yet been consistently available in schools. Schools may be the best location to equitably manage the mental health symptoms of autistic youth. In fact, youth from low-income households and/or other underserved communities are most likely to access services only in school settings. Thus, there is a critical need for evidence-based mental health interventions in schools for autistic students. The primary purpose of the current study is to compare two school-based curriculums: Facing Your Fears - Schools Based (FYF-SB) and Zones of Regulation (ZOR) on meaningful outcomes. The results of this study will not only fill a significant gap in the literature but will provide practical information about the strengths and weaknesses of each program so that school leaders and other stakeholders can make informed decisions about program selection for autistic students.

Study Aims. Aim 1: Compare the effectiveness of FYF-SB and ZOR for 200 school-aged autistic students with interfering anxiety.

Compare the effectiveness of FYF-SB and ZOR on: (a) symptoms of anxiety (primary) and emotion dysregulation (co-primary) as rated by caregivers, students, teachers, and masked research staff; and (b) functional outcomes of priority to stakeholders, including school attendance, disciplinary action, and academic participation (secondary). Hypothesis: Students who received FYF-SB will show greater reduction of anxiety compared to students who received ZOR.

Aim 2. Compare the acceptability, appropriateness, and feasibility of FYF-SB and ZOR via a mixed methods approach with students, caregivers and school providers to aid in decision-making regarding program selection (Secondary). Following intervention completion, participants will complete measures on acceptability, appropriateness, and feasibility of either FYF-SB or ZOR. In addition, a purposive subset of participants will participate in exit interviews to understand outcomes of interest, including potential harms linked with either FYF-SB or ZOR.

Aim 3. Examine autism symptom severity and anxiety symptoms severity as moderators of treatment response. This exploratory aim may help answer questions regarding which program could work best for which students.

Study Description: This study is a multi-site cluster randomized controlled, type 1 hybrid comparative effectiveness-implementation trial designed to examine whether FYF-SB or ZOR is more effective in treating anxiety in autistic students. School administrators in Colorado and North Carolina will select schools with large numbers of students from historically underserved communities. Randomization will occur at the school level to either FYF-SB (50 schools) or ZOR (50 schools). Interdisciplinary school providers (ISPs) will be trained in one of the interventions and then nominate autistic students with anxiety for participation. ISPs will deliver the intervention programs to small groups (2-5 students) in their schools. Assessments will be conducted pre, post and 6 months following program completion. Independent evaluators masked to condition will complete post-assessments. Implementation outcomes (acceptability and feasibility) will also be examined via mixed-methods and reported by students, caregivers and ISPs.

Main components of the intervention and comparator (s): The two school-based curriculums in this study are: Facing Your Fears- School Based (FYF-SB) and Zones of Regulation (ZOR). Both are rooted in CBT principles but manage anxiety in different ways. FYF-SB is based on disorder-specific CBT strategies tailored for reduction of anxiety symptoms and incorporates psychoeducation and graded exposure (facing fears a little at a time) to target anxiety. ZOR is an example of a transdiagnostic approach to intervention and targets emotion dysregulation by focusing on four different emotional states called zones. Students are taught strategies for managing emotions and how to stay in a certain zone. A transdiagnostic treatment approach posit that when emotion regulation improves so to will psychiatric symptoms related to those emotions (e.g., anxiety).

Study Population: There are three groups of participants in the study: autistic students, caregivers and interdisciplinary school providers (ISPs). (1) 200 autistic students with interfering anxiety (8-14 years) from historically underserved communities attending elementary or middle schools in Colorado or North Carolina; (2) 200 caregivers of the eligible autistic students; and (3) 150 ISPs (e.g., school psychologists, special educators, speech/language pathologists, occupational and physical therapists) who work with autistic students

Primary Outcomes: The primary outcome (s) for this study are: (1) Screening for Childhood Anxiety and Related Emotional Disorders - Child/Parent versions (SCARED; Birmaher et al. 1999). The SCARED is a 41-item inventory of statements that assesses five types of anxiety experienced by children and adolescents, to be completed separately by caregivers and students pre/post intervention and at 6 months follow-up. A total score, as well as cutoffs for specific domains of anxiety (e.g., social, generalized) are obtained. (2) Co-Primary Outcome: Pediatric Anxiety Rating Scale- Autism Spectrum Disorder (PARS-ASD) (Maddox et al. 2020). The PARS-ASD is a clinician-rated semi-structured interview assessing anxiety severity and impairment over the past week, modified for youth with ASD ages 5 to 17 from the original Pediatric Anxiety Rating Scale (PARS) (RUPP) (Walkup et al. 2013). The PARS-ASD will be administered by an independent evaluator (IE) masked to condition. It includes: a Symptom Checklist and five Severity Items.

Secondary Outcomes: There are multiple secondary outcomes: (1) stakeholder (patient-centered) identified meaningful outcomes (e.g., tardies, school attendance, grades, number of elopements, classroom participation, use of coping strategies, increase in social initiations, number of phone calls home, visits to the principal, and number of expulsions/suspensions); (2) Emotion Dysregulation Inventory (EDI) (Mazefsky et al. 2018). The EDI is a parent report measure of emotion dysregulation in youth with ASD and will be completed pre/post intervention and at follow-up. The EDI can be used as a self-report measure and can also be completed by school providers); (3) The School Anxiety Scale-Teacher Report (SAS-TR) (Lyneham et al. 2008) is a 16-item teacher-reported measure of anxiety designed to assess the behavior of children at school from 5 to 12 years of age. Items are answered on a four-point scale. The measure provides a total score for anxiety (scores ranging from 0-48); (4) Strengths and Difficulties Questionnaire (SDQ) (Goodman et al. 2000) is a 25-item teacher, parent and student reported tool measuring prosocial behavior and psychopathology of youth 3-16 years old;(5) Emotion Regulation Index for Children and Adolescents (ERICA) (MacDermott et al. 2010) is a 16-item self-report measure of social competence and emotion regulation for children between the ages of 9-16.

Implementation Outcomes: (1) CBT Program Use. This brief measure will be administered to ISPs to obtain information about their knowledge and perceptions related to school based interventions, including ZOR and FYF-SB. (2) Acceptability Questionnaire. A six-item acceptability questionnaire will be completed by students and caregivers asking them to respond to questions such as "How much did you enjoy participating in FYF-SB/ZOR?" or "My child is less anxious after participating in FYF-SB/ZOR?" A 5-point Likert scale will be used to rate their responses. (3) Implementation Survey: Brief evaluation forms using a 6-point Likert scale will be completed by ISPs post delivery of FYF-SB/ZOR to assess quality of the training, feasibility, acceptability, and appropriateness of each program including the likelihood that providers will continue to implement the interventions once the study has ended; (4) Semi-structured Exit Interviews: A purposive subset of participants (students, ISPs, caregivers) will be engaged in semi-structured exit interviews conducted by an independent member of the research team designed to understand the acceptability, appropriateness, feasibility and potential harms or negative aspects of either FYF-SB and ZOR. (5) FYF-SB/ZOR Treatment Fidelity Checklists (for internal use only). These checklists will assess ISPs' adherence to either core components of FYF-SB or ZOR, including the four ZOR key elements of preparation, provision of structure, quality of facilitation, and adult evaluation of student learning. The measures assesses the presence/absence of core treatment components as well as quality of intervention delivery.

Timeframe: Assessments occur pre and post-intervention for primary and secondary outcomes. Selected measures will also be administered at 6 months follow-up, with the 6 month follow up as primary endpoint.

Analytic Plan:

General consideration of statistical modeling: Between-arm imbalance of baseline characteristics will be examined using t and chi-square tests and evaluated based on summary statistics. Intervention effect of FYF-SB as compared to ZOR will be assessed using Linear mixed effect model (LMM) for continuous outcomes and non-linear mixed effect model (NLMM) for categorical outcome such as school attendance. To account for design effect of clustering trials, random school (cluster) effect will be in the models for outcome without repeated measures while appropriate covariance structure of LMM/NLMM accounting for both the design effect and the correlation of repeated measures will be used for outcome with repeated measures. Transformation of outcome (ie. Square root or log) will be used if normality assumption is violated. Any imbalanced potential confounding variables will be adjusted for modeling. Primary analysis will be conducted on intent-to-treat basis (ITT). LMM and NLMM will the primary method for dealing with missing value without data imputation since missing pattern would most likely be of the missing at random (MAR) pattern. The change score from baseline to the end of intervention is considered to the primary effectiveness endpoint. No type I error adjustment for multiple tests in a single model or multiple outcomes will be applied. P < 0.05 is deemed statistically significant. No interim analysis will be performed. To examine the robustness of primary analyses, sensitivity analyses will be conducted, including the same analyses among completers and analyses after missing data were imputed using Markov chain Monte Carlo (MCMC) method.

ELIGIBILITY:
Inclusion Criteria: There are 3 groups of participants: students, caregivers and interdisciplinary school providers:

Inclusion criteria for students ages 8-14:

* known medical diagnosis of ASD OR educational identification of ASD OR suspected ASD
* clinical anxiety according to either student, parent or teacher report
* clinically significant impairment (T-score above 70) in reciprocal social behavior according to the Social Responsiveness Scale - Second Edition (SRS-2).

Exclusion criteria for students

* known intellectual disability
* significant behavior or psychiatric challenge that prevents them from participation in small group activities
* lack of parent or caregiver permission for participation

Inclusion Criteria for Caregivers of students 8-14

- legal guardian of a student who meets inclusion criteria defined above

Inclusion criteria for Interdisciplinary school providers (ISPs).

* degreed professionals in one of the following: education (special or general education), school psychology, counseling, social work, speech/language pathology, occupational or physical therapy OR paraprofessional who assist ISPs
* working with autistic students with anxiety
* be able to complete study requirements including attending the training workshops, delivering at least 80% of the program they were randomized to, and participating in 80% of bi-monthly consultation sessions with the research team.

Exclusion criteria ISPs

* if they are unable to participate in the trainings, deliver the program they are assigned to, or participate in any of the consultation visits
* if they do not work with students with autism and anxiety

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in anxiety on the clinician-administered Pediatric Anxiety Rating Scale - Autism Spectrum Disorder (PARS-ASD) | Baseline, within 4 weeks post-intervention; and 6 months after completion of the intervention
  The PARS-ASD is a clinician administered semi-structured interview to assess anxiety symptoms and severity. The PARS-ASD will be administered by an independent evaluator (IE) masked to condition. It includes: a Symptom Checklist and five Severity Items. The Symptom Checklist covers social anxiety, separation anxiety, generalized anxiety, panic, specific phobia, and other anxiety symptoms. The severity of symptoms is examined by assessing the frequency and pervasiveness of anxiety, as well as the extent to which the child avoids anxiety provoking situations (e.g., behavioral manifestations of anxiety).
Change from Baseline in parent reported anxiety on the Screening for Childhood Anxiety and Related Emotional Disorders (SCARED) | baseline, within 4 weeks post-intervention; and 6 months after completion of the intervention
  The SCARED is a 41-item inventory of statements that assesses five types of anxiety experienced by children and adolescents, to be completed separately by caregivers and students. A total score, as well as cutoffs for specific domains of anxiety (e.g., social, generalized) are obtained. A total score of 25 or higher is clinically significant. Scores range from 0-82 and higher scores indicate a worse outcome.
Change from Baseline in child reported anxiety on the Screening for Childhood Anxiety and Related Emotional Disorders (SCARED) | baseline, within 4 weeks post-intervention; and 6 months after completion of the intervention
  The SCARED is a 41-item inventory of statements that assesses five types of anxiety experienced by children and adolescents, to be completed separately by caregivers and students. A total score, as well as cutoffs for specific domains of anxiety (e.g., social, generalized) are obtained. A total score of 25 or higher is clinically significant. Scores range from 0-82 and higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
Change from Baseline in parent reported emotion regulation and reactivity on the Emotion Dysregulation Inventory (EDI) | baseline, within 4 weeks post-intervention; and 6 months after completion of the intervention
  The EDI is a measure of emotion dysregulation in youth with ASD. The EDI can be used as a self-report measure and can also be completed by school providers. Items are rated on a 5-point Likert scale ranging from 1 (not at all) to 5 (very severe). Scores range from 0-52, and higher scores indicate a worse outcome.
Change from Baseline in child reported emotion regulation and reactivity on the Emotion Dysregulation Inventory (EDI) | baseline, within 4 weeks post-intervention; and 6 months after completion of the intervention
  The EDI is a measure of emotion dysregulation in youth with ASD. The EDI can be used as a self-report measure and can also be completed by school providers. Items are rated on a 5-point Likert scale ranging from 1 (not at all) to 5 (very severe). Scores range from 0-52, and higher scores indicate a worse outcome.
Change from Baseline in teacher reported emotion regulation and reactivity on the Emotion Dysregulation Inventory (EDI) | baseline, within 4 weeks post-intervention; and 6 months after completion of the intervention
  The EDI is a measure of emotion dysregulation in youth with ASD. The EDI can be used as a self-report measure and can also be completed by school providers. Items are rated on a 5-point Likert scale ranging from 1 (not at all) to 5 (very severe). Scores range from 0-52, and higher scores indicate a worse outcome.
Change from Baseline in teacher reported anxiety on The School Anxiety Scale - Teacher Report (SAS-TR) | baseline, within 4 weeks post-intervention; and 6 months after completion of the intervention
  The SAS-TR is a 16-item teacher-reported measure of anxiety designed to assess the behavior of children at school. Items are answered on a four-point scale. The measure provides a total score for anxiety (scores ranging from 0-48; higher score indicate a worse outcome). It includes two subscale scores (reflecting social anxiety and generalized anxiety).
Change from Baseline in child reported social competence and emotion regulation on the Emotion Regulation Index for Children and Adolescents (ERICA) | baseline, within 4 weeks post-intervention and 6 months after completion of the intervention
  ERICA is a 16-item self-report measure of social competence and emotion regulation for children between the ages of 9-16. Students use a 5-point Likert scale to respond to the items. ERICA measures three factors: emotional control, emotional self-awareness, and situational responsiveness. Scores range from 16-80, and higher scores indicate a worse outcome.
Change from Baseline in parent reported prosocial behavior and psychopathology on the Strengths and Difficulties Questionnaire (SDQ). | baseline, within 4 weeks post-intervention and 6 months after completion of the intervention
  SDQ is a 25-item teacher, parent and student reported tool measuring prosocial behavior and psychopathology of youth 3-16 years old. The SDQ evaluates five-factors: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. Scores range from 0-50 with higher scores indicating better outcomes.
Change from Baseline in child reported prosocial behavior and psychopathology on the Strengths and Difficulties Questionnaire (SDQ). | baseline, within 4 weeks post-intervention and 6 months after completion of the intervention
  SDQ is a 25-item teacher, parent and student reported tool measuring prosocial behavior and psychopathology of youth 3-16 years old. The SDQ evaluates five-factors: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. Scores range from 0-50 with higher scores indicating better outcomes.
Change from Baseline in teacher reported prosocial behavior and psychopathology on the Strengths and Difficulties Questionnaire (SDQ). | baseline, within 4 weeks post-intervention and 6 months after completion of the intervention
  SDQ is a 25-item teacher, parent and student reported tool measuring prosocial behavior and psychopathology of youth 3-16 years old. The SDQ evaluates five-factors: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. Scores range from 0-50 with higher scores representing better outcomes.

OTHER OUTCOMES:
Treatment Fidelity | From the beginning of the intervention through the end of intervention, up to a period of 20 weeks, the fidelity measure will be completed weekly by the independent research team
  Independent research team will code treatment fidelity for Zones of Regulation and Facing Your Fears-School Based program
Acceptability - Children | within 4 weeks post-intervention
  A six-item acceptability questionnaire will be completed by children asking them to respond to questions such as "How much did you enjoy participating in FYF-SB/ZOR?" A 5-point Likert scale will be used to rate their responses. Scores range from 5-25 with higher scores indicating a better outcome.
Acceptability - parents | within 4 weeks post-intervention
  A six-item acceptability questionnaire will be completed by parents asking them to respond to questions such as "My child is less anxious after participating in FYF-SB/ZOR?" A 5-point Likert scale will be used to rate their responses. Scores range from 5-25 with higher scores indicating a better outcome.
Semi-structured exit interviews - Students | within 4 weeks post-intervention
  approximately 50% of students will participate in 20-30 minute interviews regarding the programs (either Zones of Regulation or Facing Your Fears).
Semi-structured exit interviews - parents | within 4 weeks post-intervention
  approximately 50% of parents will participate in 20-30 minute interviews regarding the programs (either Zones of Regulation or Facing Your Fears).
Semi-structured exit interviews - ISPs | within 4 weeks post-intervention
  approximately 50% of ISPs will participate in 20-30 minute interviews regarding the programs (either Zones of Regulation or Facing Your Fears).

CONTACTS AND LOCATIONS:
Overall Officials: Judy Reaven, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pickard K, Maddox B, Boles R, Reaven J. A cluster randomized controlled trial comparing the effectiveness of two school-based interventions for autistic youth with anxiety. BMC Psychiatry. 2024 Jan 2;24(1):6. doi: 10.1186/s12888-023-05441-0. PMID 38166851